CLINICAL TRIAL: NCT06540430
Title: Digital Based Home Care Service for Ostomy Patients: Randomized Controlled Trials
Brief Title: Digital Based Home Care Service for Ostomy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: The Korean Society of Coloproctology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ostocare2024
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Neoplasms; Stoma Colostomy; Stoma Ileostomy
Keywords: Stoma; Colorectal neoplasms; Quality of life
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention group will use a mobile application where patients input their stoma condition, allowing healthcare professionals to monitor and manage their care.
  The control group consists of patients who received conventional outpatient-based stoma care without using the application service.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App group (Experimental): The intervention group will use a mobile application where patients input their stoma condition, allowing healthcare professionals to monitor and manage their care.
  Interventions: Behavioral: The Use of a Mobile Application for Stoma Self-Care
- Conventional group (No Intervention): The control group consists of patients who received conventional outpatient-based stoma care without using the application service.

INTERVENTIONS:
Behavioral: The Use of a Mobile Application for Stoma Self-Care — The intervention group will use a mobile application where patients input their stoma condition, allowing healthcare professionals to monitor and manage their care. The app provides patients with information on diet, physical activity, stoma care, emotional support, and daily living needs.
  Arms: App group

SUMMARY:
This study aims to enhance the physical, psychological, and social aspects of stoma care by providing a self-management service via a smartphone application, and to evaluate the impact of this digital-based application on patients' quality of life.

DETAILED DESCRIPTION:
This study will include patients who have undergone colorectal cancer surgery and received either a colostomy or ileostomy, provided they are comfortable using digital devices like smartphones. Patients will be randomly assigned to either the intervention group, receiving stoma care through a smartphone application, or the conventional group, receiving standard outpatient-based care. The intervention group will use a mobile application where patients input their stoma condition, allowing healthcare professionals to monitor and manage their care. The app provides patients with information on diet, physical activity, stoma care, emotional support, and daily living needs. Both groups will be assessed for outcomes at the time of enrollment, and at 1 and 6 months. Outcome measures include stoma-related complications such as peristomal dermatitis, dehydration, acute renal failure, readmission due to stoma-related issues, and quality of life and emotional state assessments using EQ-5D-5L and Stoma Quality of Life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years or older
* Patients who have a colostomy or ileostomy after surgery for colon cancer
* Patients who do not have difficulty using a smartphone

Exclusion Criteria:

* Patients younger than 19 years
* Patients aged 80 years or older
* Patients who do not know how to use a smartphone
* Patients with cognitive impairments
* Patients with pre-existing psychiatric disorders
* Patients who have undergone emergency surgery
* Patients who already have stoma-related complications

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Peristomal Dermatitis | enrollment, 1 month, and 6 months.
  Evaluated using the DET Score (Discoloration, Erosion, and Tissue Overgrowth) on a scale ranging from 0 to 3.
Wound Infection, stoma retraction, bleeding, hernia, and Acute kidney injury | enrollment, 1 month, and 6 months.
  Incidence rate as a percentage of patients affected.
Readmission Rate | enrollment, 1 month, and 6 months.
  Incidence rate as the percentage of patients readmitted due to stoma-related complications.

SECONDARY OUTCOMES:
Evaluation of Anxiety and Depression | enrollment, 1 month, and 6 months.
  The EuroQol-5 Dimension (EQ-5D) will be utilized to gauge the general health status.
  The EQ-5D-5L score consists of two components. One component is the Visual Analogue Scale (VAS), which assesses an individual's overall health status on a scale from 0 to 100. A score of 0 represents "the worst imaginable health state," while a score of 100 represents "the best imaginable health state." The other component assesses health status across five dimensions, each rated on a five-level scale ranging from 1 (no problems) to 5 (extreme problems). The combination of these five dimensions represents a specific health state, and a value set specific to each country is used to calculate a score based on this state. This score typically ranges from 0 to 1, with 1 indicating "perfect health."
Evaluation of Quality of Life | enrollment, 1 month, and 6 months.
  The Stoma Quality-of-Life Scale will be used to assess the quality of life specifically related to stoma management and its impacts.
  The Stoma-QoL questionnaire consists of 20 questions, with a total score range from 20 to 80. Higher scores indicate a better quality of lif

IPD SHARING:
Plan to Share IPD: Undecided